CLINICAL TRIAL: NCT00621894
Title: A Phase IIA Randomized, Double-Blind, Placebo-Controlled Study of LGD-4665 in Patients With Immune Thrombocytopenic Purpura (ITP) With an Open Label Extension
Brief Title: Oral LGD-4665 Versus Placebo in Adults With Immune Thrombocytopenic Purpura (ITP) for 6 Weeks Plus Open Treatment Continuation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L4665-03
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Immune thrombocytopenic purpura; thrombopoietin mimetic; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LGD4665 (Experimental): LGD-4665: Experimental Thrombopoietin mimetic
  Interventions: Drug: LGD-4665
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LGD-4665 — LGD-4665 Thrombopoietin mimetic
  Arms: LGD4665
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the ability of LGD-4665 given daily by mouth to increase platelet counts in the treatment of patients with ITP (immune thrombocytopenic purpura). LGD-4665 increased platelet counts safely and tolerably compared to placebo in healthy volunteers. This study will examine the safety, tolerability and efficacy of 7.5 mg capsules of LGD-4665 to increase platelets compared to placebo, randomized 2:1, during blinded treatment for 6 weeks. Evaluation of platelet counts, bleeding scores and safety parameters will be done weekly. All patients are eligible to continue on active, open LGD-4665 treatment for an additional 12 weeks with optimal adjustment of dose for each patient.

DETAILED DESCRIPTION:
This is a Phase IIA study with two parts to the design.

* Part 1 is a randomized, double-blinded, placebo-controlled treatment of 7.5 mg/day LGD-4665 versus placebo in approximately 24 patients with ITP who have been treated with at least one prior therapy for ITP. Patients will be randomized in a ratio of 1:2 (placebo: 7.5 mg/day LGD-4665) for 6 weeks of treatment. Platelet counts, bleeding scores, vital signs, physical exams and laboratory tests will be assessed weekly. Treatment groups will be analyzed for efficacy by the percentage of patients with platelet counts two times baseline and ≥ 50,000/uL at 6 weeks of treatment, and for safety by adverse events, vital signs, physical exams, laboratory tests and use of ITP rescue medications or transfusions.
* Part 2 is an extension of study treatment with open label LGD-4665. All patients who participate in the Part 1 randomized double-blind treatment of this Ph IIA trial are eligible to continue open label treatment with LGD-4665 for up to 3 months at an appropriate dose for the safe maintenance of platelet counts (≥ 50,000/uL to ≤ 200,000/uL). Assessments of effectiveness and safety will be made at 2 and 4 week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Diagnosis of ITP for at least 3 months consistent with ASH guidelines
* Treated with one or more prior therapies for ITP and platelet counts < 30,000/µL or < 50,000/µL if on a stable oral corticosteroid for ≥ 4 weeks, supported by 2 platelet counts in prior 30 days
* Laboratory results within normal range except for the following analytes

  * Hemoglobin ≥ 10 g/dL
  * Absolute neutrophil counts > 1000/mL
  * ALT ≤ 1.5X ULN
  * AST ≤ 1.5X ULN
  * Creatinine < 1.5X ULN
  * Bilirubin < 1.5X ULN
  * BUN < 1.5X ULN
  * PT < 1.5X ULN
  * aPTT <1.5X ULN
* Women of child-bearing potential must have a negative serum pregnancy test within 4 days prior to the first dose of study treatment and agree to practice an approved method of contraception or abstinence from sexual intercourse.
* Willing to sign a written informed consent

Exclusion criteria:

* History of heart attack or cardiovascular disease
* Known history of arterial or venous thrombosis
* More than 3 risk factors for thromboembolic events (diabetes, smoker, using oral contraception, using estrogen therapy, hypertriglyceridemia, average cholesterol > 240 mg/dL, treatment for hypertension)
* Active cancer or a history of bone marrow disorders
* Women who are pregnant or nursing
* History of alcohol/drug abuse or dependence within one year
* Listed medications dosed within:

  * 4 weeks of the first dose of the study treatment:

    * Use of Rituximab
    * Use of cytotoxic agents
    * Use of Cyclosporine and other immunomodulators
    * Use of an investigational drug
  * 2 weeks of the first dose of the study treatment:

    * Use of Danazol
    * Use of Azathioprine
    * Use of Mycophenolate mofetil and pulsed-dose steroids
  * 1 week of the first dose of the study treatment:

    * Use of Anti-D (WinRho®)
    * Use of IVIG
    * Had a platelet transfusion
    * Use of herbal/dietary supplements (excluding vitamins and mineral supplements)
  * 3 days of the first dose of the study treatment

    * Use of aspirin, aspirin containing compounds
    * salicylates
    * milk of magnesia
    * non-steroidal anti-inflammatory drugs (unless prescribed for heart disease)
* History of platelet aggregation that would prevent measurement of platelet counts
* Known active infection with HIV, hepatitis B, or hepatitis C
* In the Investigator's opinion, the patient is not able to comply with requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-03-15 (Actual); Primary Completion 2009-05-01 (Actual); Study Completion 2009-05-15 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with platelet count >= 50000/µL | At Week 6
  Response was defined as platelet count >= 50 x1000/uL for participants without Baseline steroid uses; or platelet counts >= 50 x1000/uL and doubling the Baseline platelet counts for participants with baseline steroid uses. Confidence interval of response rate was computed using exact method of binomial proportion.

SECONDARY OUTCOMES:
Number of participants with time to response by Platelet Counts (platelet counts >= 50,000/µL) | Week 1, 2, 4 and 6 of part 1
  Response was defined as platelet count >= 50 x1000/uL for participants without baseline steroid uses; or platelet counts >= 50 x1000/uL and doubling the Baseline platelet counts for participants with baseline steroid uses.
Change From Baseline to Last Bleeding Observation During Double-Blind Treatment | Day 1 (Baseline) and Week 6
  ITP Bleeding Severity Scale was used for the analysis of bleeding score. Bleeding scores were, 0=None, 1=minor, and 2=major. Body sites and bleeding grade analysis was as follows: cutaneous (1= 1-5 bruises; scattered petechiae and 2= > 5 bruises, >2 centimeter [cm]; petechiae), oral mucosa (1= 1 blood blister or > 5 petechiae, gum bleeding < 5 minute[min], 2= multiple blood blisters; gum bleeding > 5 min), epistaxis (1= blood on blowing nose or epistaxis < 5 min, 2= bleeding > 5 min), gastrointestinal (1= occult blood, 2= gross blood), gynecological (1= spotting not at time of period, 2= bleeding not at time of period or very heavy period), urinary (1= microscopic (+ by dipstick), 2= macroscopic), pulmonary(1= possible symptoms but mild, 2= yes), subconjunctival (1= yes, 2= both eyes significantly involved), Intracranial (1= possible symptoms, 2= yes, clinically confirmed). Change from Baseline was calculated as Baseline value minus post-randomization value. Baseline was Day 1value.
Duration of platelet counts >= 50,000/µL of LGD4665 | Up to Week 6
  Response was defined as platelet count >= 50 x1000/uL for participants without baseline steroid uses; or platelet counts >= 50 x1000/uL and doubling the Baseline platelet counts.A Kaplan-Meier projection of time to response by platelet counts was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (15):
  - University of California San Diego Medical Center, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Davis, Posteraro and Wasser, MD's LLP, Manchester, Connecticut
  - Baptist Cancer Institute, Jacksonville, Florida
  - Cancer Center of Florida, Orlando, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Karmanos Cancer Center, Wertz Clinical Cancer Center 4HWCRC, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine - St Louis, MO, St Louis, Missouri
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Joan and Sanford I. Weill Medical College, Cornell University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Case Western Reserve University School of Medicine, Cleveland, Ohio
  - Cleveland Clinic Foundation, Univ. of Ohio, Cleveland, Ohio
  - Hematology Oncology Associates of South Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

REFERENCES:
- See also: Results for study L4665-03 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/L4665-03?search=study&search_terms=L4665-03#rs